CLINICAL TRIAL: NCT06610669
Title: The Prevalence, Patients' Characteristics, and Hyper-Lp(a)-Emia Risk Factors in the Polish Population. The Polish Mother's Memorial Hospital Research Institute Lipoprotein(a) Registry
Brief Title: The Prevalence of Hyper-Lp(a)-Emia in the PMMHRI-Lp(a) Registry
Status: Recruiting | Type: Observational
Sponsor: Polish Mother Memorial Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PMMHRI-Lp(a)-Registry
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-08

CONDITIONS: Lipoprotein(a), Hyper-Lp(a)-Emia
Keywords: lipoprotein(a)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The PMMHRI-Lp(a)-Registry is a non-interventional, single-center registry conducted in the Polish Mother's Memorial Hospital Research Institute (PMMHRI). The PMMHRI-Lp(a)-Registry was established in January 2022. Since then, all consecutive patients of the Department of Cardiology and Adult Congenital Heart Diseases, Department of Endocrinology, and outpatient cardiology and endocrinology clinics with the measured Lp(a) concentration have been included.

DETAILED DESCRIPTION:
The PMMHRI-Lp(a)-Registry is a non-interventional, single-center registry conducted in Poland's 2nd largest, supra-regional hospital - the Polish Mother's Memorial Hospital Research Institute (PMMHRI). The PMMHRI-Lp(a)-Registry was established in January 2022. Since then, all consecutive patients of the Departments of Cardiology, Endocrinology, and outpatient cardiology and endocrinology clinics have been included. The indications for Lp(a) measurement in the registry are based on the 2021 Polish Lipid Guidelines and new Polish recommendations on the management of elevated Lp(a) (2024). Lp(a) was determined using Sentinel's Lp(a) Ultra, an Immunoturbidimetric quantitative test (Sentinel, Milan, Italy), and the results are presented in mg/dl.

The following information was collected from the patient's medical records: demographic parameters; relevant comorbidities; concomitant medications including lipid-lowering therapy status, anticoagulation status; smoking status; post hoc calculated cardiovascular risk score; and laboratory parameters including i.e. Lp(a) and lipids profile.

ELIGIBILITY:
Inclusion Criteria:

* measured lipoprotein(a) concentration

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients of the Department of Cardiology and Adult Congenital Heart Diseases, Department of Endocrinology, and outpatient cardiology and endocrinology clinics with the measured Lp(a) concentration.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Prevalence of hyper-Lp(a)-aemia among the Polish population, along with the identification of associated patient characteristics and risk factors | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Polish Mother Memorial Research Institute, Lodz, Poland